CLINICAL TRIAL: NCT04341285
Title: Early Versus Late ECMO Therapy in COVID-19 Induced ARDS (ECMO-VID)
Acronym: ECMO-VID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study protocol was changed to include non-COVID patients and registered under a different ID
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Freiburg (Other); RWTH Aachen University (Other); University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECMO-VID
Record Dates: First submitted 2020-03-30; First posted 2020-04-10 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2020-06

CONDITIONS: ARDS, Human; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Experimental intervention: Insertion of Extracorporal Membrane Oxygenation (ECMO) within 24 hours Control intervention: Insertion of Extracorporal Membrane Oxygenation (ECMO) as rescue therapy following failure of conventional therapy for ARDS. This conventional therapy will be standardized to reduce bias.
  Duration of intervention per patient: varies, depending on severity of pulmonary compromise Follow-up per patient: 90days or until hospital discharge Accompanying measures: Serum Samples and bronchoscopy samples of patients included into the trial for secondary analysis of inflammatory parameters and potential biomarkers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early ECMO (Active Comparator): Experimental intervention: Insertion of Extracorporal Membrane Oxygenation (ECMO) within 24 hours of referral to an Intensive Care Unit.
  Interventions: Procedure: ECMO Implantation
- Late ECMO (Active Comparator): Insertion of Extracorporal Membrane Oxygenation (ECMO) as rescue therapy following failure of conventional therapy for ARDS. This conventional therapy will be standardized to reduce bias.
  Interventions: Procedure: ECMO Implantation

INTERVENTIONS:
Procedure: ECMO Implantation — Insertion of Extracorporal Membrane Oxygenation (ECMO) within 24 hours of referral to an Intensive Care Unit.

SUMMARY:
Experimental intervention: Insertion of Extracorporal Membrane Oxygenation (ECMO) within 24 hours of referral to an Intensive Care Unit.

Control intervention: Insertion of Extracorporal Membrane Oxygenation (ECMO) as rescue therapy following failure of conventional therapy for ARDS. This conventional therapy will be standardized to reduce bias.

Duration of intervention per patient: varies, depending on severity of pulmonary compromise Follow-up per patient: Until hospital discharge Accompanying measures: Serum Samples and bronchoscopy samples of patients included into the trial for secondary analysis of inflammatory parameters and potential biomarkers

DETAILED DESCRIPTION:
The severe form of COVID-19 infection is characterized and marked by severe pneumonia and the Acute Respiratory Distress Syndrome (ARDS). ARDS is characterized by the loss of pulmonary tissue compliance and severe hypoxia. The central pathophysiologic changes of COVID-19+ ARDS are dysregulated inflammation within the alveolar space and altered permeability of the alveolar-capillary barrier. The public health impact of this COVID-19+ ARDS is considerable with a large number of ARDS cases that need to be treated currently on German Intensive Care Units. To date, the associated mortality ranges between 30 to 50%. In the ongoing COVID-19 crisis cases of ARDS will still increase and pose a significant challenge to the German Medical System. Despite the emerging understanding of COVID-19+ ARDS, treatment only remains to be symptomatic using mechanical ventilation, prone positioning and in severe cases of hypoxia extracorporal membrane oxygenation (ECMO). Current evidence generated by clinical trials demonstrates that patients with ARDS should be referred to a specialized center to receive expert treatment. The use of ECMO might have a beneficial effect on overall patient outcome, yet this has not been proven by clinical trials and to date ECMO is recommended as measure of last resort in the current ARDS treatment guidelines. The timing of ECMO placement to relieve hypoxia is an important question for the treating clinician but is not well studied to date. This might also have impact on the long-term functional outcome of patients. In addition, evidence about the role of ECMO in the outcome of COVID-19+ patients might have significant impact on the referral of patients to a specialized center and is important for the treating physician. Therefore, the investigators want to pursue the questions whether early ECMO placement is superior than the placement of ECMO as a rescue measure, and whether this could result in improved overall outcome of patients with COVID-19+ ARDS.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19positive(+) ARDS as defined according to the Berlin Definition
* ratio of partial pressure arterial oxygen and fraction of inspired oxygen (PaO2/ FiO2) ≤100
* Bilateral opacities consistent with pulmonary edema on frontal chest radiograph
* requirement for positive pressure ventilation via an endotracheal tube or non-invasive ventilation
* no clinical evidence of left atrial hypertension, or if measured, a Pulmonary Arterial Wedge Pressure (PAOP) less than or equal to 18 mmHg.
* ≤ 7 days from the initiation of mechanical ventilation at the time of randomization. - Patients must be enrolled within 96 hours of onset of ARDS -

Exclusion Criteria:

* COVID-19negative(-) ARDS
* Age less than 18 years
* More than 7 days since initiation of mechanical ventilation
* more than 96 hours since meeting ARDS criteria
* patient, surrogate or physician not committed to full intensive care support.
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
28 day all cause mortality | 28 Days
  survival in 28-day follow-up period (28 day all cause mortality)

SECONDARY OUTCOMES:
90 day all cause mortality | 90 days
  90 day all cause mortality
Sepsis-related organ failure assessment score at day 1-14, 28 and 90 days | day 1-14, 28 and 90
  Sepsis-related organ failure assessment score at day 1-14, 28 and 90 days
duration of mechanical ventilation support | 28 days
  duration of mechanical ventilation support
Ventilator Associated Pneumonia | 28 days
  Number of patients with Ventilator Associated Pneumonia
Bleeding complications | 28 das
  number of blood transfusion units
Acute Renal Failure | 28 days
  Days on real replacement therapy
Discharge Location | 90 days
  Discharge to (home, skilled nursing facility, rehabilitation)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenberger, Prof., Principal Investigator — +4970712986622
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided